CLINICAL TRIAL: NCT02801448
Title: Randomized Clinical Trial With Broccoli Sprout Extract to Patients With Type 2 Diabetes
Brief Title: Clinical Trial With Broccoli Sprout Extract to Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anders Rosengren, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Anders Rosengren, MD PhD, MD PhD, Region Skane
Organization: Region Skane (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BSE1
Record Dates: First submitted 2016-06-12; First posted 2016-06-15 (Estimated); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — sulforaphane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo containing maltodextrine but no active sulforaphane
  Interventions: Drug: Placebo
- BSE (Active Comparator): Broccoli sprout extract once daily for 12 weeks
  Interventions: Drug: sulforaphane

INTERVENTIONS:
Drug: sulforaphane — sulforaphane-containing broccoli sprout extracts
  Arms: BSE
Drug: Placebo — Maltodextrine-based placebo without sulforaphane
  Arms: Placebo

SUMMARY:
Type 2 diabetes (T2D) results from a combination of insufficient insulin secretion from pancreatic islets and insulin resistance of target cells. The investigators have extensive pre-clinical data suggesting that BSE through its high content of the isothiocyanate sulforaphane improves hepatic insulin sensitivity. BSE as a dietary supplement could therefore benefit both patients with T2D and individuals at risk for the disease. BSE-containing sulforaphane is suggested to activate Nuclear factor-like 2 (NRF2). The investigators aim to study the clinical effect of using BSE as a dietary supplement on glucose tolerance and insulin sensitivity.

DETAILED DESCRIPTION:
Sulforaphane binds to Keap1 in the cytosol, leading to nuclear translocation of this transcription factor. In the nucleus NRF2 induces the expression of a large number of anti-oxidative genes. Sulforaphane is contained at high concentration in broccoli sprout extracts (BSE). Human studies have been conducted using broccoli sprout products without complication. It is being tested for the treatment or prevention of cancer and inflammatory diseases in ~30 clinical trials without any serious adverse events reported. The low toxicity makes BSE ideal as a dietary supplement for preventing and treating T2D.

The investigators aim to study the clinical effect of sulforaphane on glucose tolerance in T2D patients. Sulforaphane will be given as BSE. BSE is a freeze-dried powder of an aqueous extract of broccoli sprouts that provides a consistent and stable source of sulforaphane. The investigators will use a parallel arm study design with patients receiving BSE or placebo. The randomization will be double-blind. The study will be done at one centre. Patients with BMI between 25-40 kg/m2 will be included. Another inclusion criterion is HbA1c 6-10%. Patients will be treated for 12 weeks to enable us to observe effects on HbA1c (HbA1c turn-over is 3 months).

Patients will come to a screening visit and if they give informed consent and are included they attend a second visit 2-3 weeks later.

The patients will undergo an oral glucose tolerance test (OGTT) before and after the 12-week treatment period. The reason for using OGTT rather than e.g. insulin clamps as the readout is that it is a harmless standard procedure that gives an integrated view of glucose tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Classified as type 2 diabetes
* Written informed consent
* Age: for men and women 35-75 years; for women below 75 years should be postmenopausal (defined as no menstrual bleeding since at least one year).
* Body mass index 25-40 kg/m2
* At screening visit : HbA1c 6-10 %, equivalent to 41-86 mmol/mol
* Currently treated with metformin or diet

Exclusion Criteria:

* Treatment with insulin, other anti-diabetic treatment given as injections or any oral anti-diabetic treatment except metformin
* Fasting blood glucose at screening > 15.0 mmol/L
* Active liver disease
* At screening or at any subsequent visit a level of aspartate aminotransferase (ASAT) or alanine aminotransferase (ALAT) of more than three times the upper limit of the normal range
* Gastrointestinal ailments which may interfere with the ability to adequately absorb sulforaphane
* At screening visit creatinine > 130 µmol/L
* Coagulation disorder or current anti-coagulant therapy with warfarin, which may be affected by the BSE
* Diagnosed with a cardiovascular disease or event within 6 months prior to enrolment
* Systemic glucocorticoid treatment
* Herbal treatment, defined as food supplement (except multivitamin treatment) with herbal or vegetable extracts that may contain sulforaphane
* Allergy to broccoli
* Mental disorder making the patient unable to understand the study information
* Participation in other clinical trial which may affect the outcome of the present study
* Any other physical or psychiatric condition or treatment that in the judgment of the investigator makes it difficult to participate in the study.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2015-09; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Delta-HbA1c | 12 weeks
  difference in HbA1c before and after treatment

SECONDARY OUTCOMES:
Delta-fasting blood glucose | 12 weeks
  difference in fasting blood glucose before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anders Rosengren, Principal Investigator — Lund University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Axelsson AS, Tubbs E, Mecham B, Chacko S, Nenonen HA, Tang Y, Fahey JW, Derry JMJ, Wollheim CB, Wierup N, Haymond MW, Friend SH, Mulder H, Rosengren AH. Sulforaphane reduces hepatic glucose production and improves glucose control in patients with type 2 diabetes. Sci Transl Med. 2017 Jun 14;9(394):eaah4477. doi: 10.1126/scitranslmed.aah4477. PMID 28615356